CLINICAL TRIAL: NCT04225871
Title: A Phase 3, Multicenter, Open-Label Extension Study of Zilucoplan in Subjects With Generalized Myasthenia Gravis
Brief Title: Open-Label Extension of Zilucoplan in Subjects With Generalized Myasthenia Gravis
Acronym: RAISE-XT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA101495-02.302; 2024-512399-37 (Registry Identifier: EU Clinical Trials); U1111-1306-6625 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-10-02; First posted 2020-01-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — zilucoplan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 0.3 mg/kg zilucoplan (RA101495) (Experimental)
  Interventions: Drug: zilucoplan (RA101495)

INTERVENTIONS:
Drug: zilucoplan (RA101495) — Daily subcutaneous (SC) injection

SUMMARY:
The RAISE-XT study is an open-label extension study to evaluate the long-term efficacy, safety, and tolerability of zilucoplan in subjects with gMG who have previously participated in a qualifying Ra Pharmaceuticals sponsored zilucoplan study.

ELIGIBILITY:
Inclusion Criteria:

* Completion of a qualifying zilucoplan study

Exclusion Criteria:

* With the exception of a prior zilucoplan trial, participation in another concurrent clinical trial involving an experimental therapeutic intervention (participation in observational studies and/or registry studies is permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From Baseline (Day 1) to Safety Follow-Up Visit (up to 36 months)
  A treatment-emergent adverse event is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication.

SECONDARY OUTCOMES:
Change from Baseline to Week 12 in the Myasthenia Gravis-Activities of Daily Living (MG-ADL) Score | From Baseline (Day 1) to Week 12
  The MG-ADL profile provides an assessment of MG symptom severity and measures 8 items on a 0-3 scale, with 0 being the least severe. The total sum of the 8 items represents the ADL score. The ADL score can range from 0 (least severe) to 24 (most severe).
Change from Baseline to Week 12 in the the Quantitative Myasthenia Gravis (QMG) Score | From Baseline (Day 1) to Week 12
  The QMG test is a standardized quantitative strength scoring system and measures 13 items on a 0-3 scale, with 0 being the least severe. The total sum of the 13 items represents the QMG score. The QMG score can range from 0 (least severe) to 39 (most severe).
Change from Baseline to Week 12 in the Myasthenia Gravis Composite (MGC) Score | From Baseline (Day 1) to Week 12
  The MGC is a 10-item scale that has been used to measure the clinical status of patients with Myasthenia Gravis (MG) in order to evaluate treatment response. The MGC has 4-point Likerttype Scale response options ranging from 0 to 2, 3, 4, 5, 6 or 9 according to the item (weighted response options). The total score is the sum of all items (range 0-50) where higher scores indicate more severe impairment due to the disease.
Change from Baseline to Week 12 in the Myasthenia Gravis - Quality of Life revised (MG-QOL15r) Score | From Baseline (Day 1) to Week 12
  The MG-QOL15r is a 15-item survey that was designed to assess quality of life in patients with MG. The MG-QoL has 3-point Likert Scale response options ranging from 0 to 2. The MGQoL15r score can range from 0 to 30, where higher scores indicate more severe impact of the disease on aspects of the patient's life.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (70):
- United States (33):
  - Mg0011 41, Mobile, Alabama
  - Mg0011 116, Phoenix, Arizona
  - Mg0011 31, Irvine, California
  - MG0011 4, Los Angeles, California
  - Mg0011 220, Pasadena, California
  - Mg0011 160, San Francisco, California
  - Mg0011 24, New Haven, Connecticut
  - Mg0011 27, Washington D.C., District of Columbia
  - Mg0011 25, Tampa, Florida
  - Mg0011 135, Augusta, Georgia
  - Mg0011 188, Glenview, Illinois
  - Mg0011 156, Indianapolis, Indiana
  - Mg0011 32, Kansas City, Kansas
  - Mg0011 33, Detroit, Michigan
  - Mg0011 49, East Lansing, Michigan
  - Mg0011 134, Columbia, Missouri
  - Mg0011 117, Las Vegas, Nevada
  - Mg0011 30, Buffalo, New York
  - Mg0011 123, Great Neck, New York
  - Mg0011 23, New York, New York
  - Mg0011 47, New York, New York
  - Mg0011 22, Chapel Hill, North Carolina
  - Mg0011 122, Cleveland, Ohio
  - Mg0011 38, Columbus, Ohio
  - Mg0011 40, Pittsburgh, Pennsylvania
  - Mg0011 128, Charleston, South Carolina
  - Mg0011 28, Cordova, Tennessee
  - Mg0011 131, Austin, Texas
  - Mg0011 19, Dallas, Texas
  - Mg0011 39, Salt Lake City, Utah
  - Mg0011 164, Charlottesville, Virginia
  - Mg0011 154, Seattle, Washington
  - Mg0011 45, Milwaukee, Wisconsin
- Mg0011 11, Montreal, Canada
- France (4):
  - Mg0011 204, Lille
  - Mg0011 118, Nice
  - Mg0011 105, Paris
  - Mg0011 137, Strasbourg
- Germany (2):
  - Mg0011 150, Göttingen
  - Mg0011 129, Tübingen
- Italy (2):
  - Mg0011 132, Milan
  - Mg0011 126, Roma
- Japan (10):
  - Mg0011 151, Chiba
  - Mg0011 136, Hanamaki-shi
  - Mg0011 179, Kita-gun
  - Mg0011 153, Meguro-ku
  - Mg0011 146, Nagasaki
  - Mg0011 169, Narita
  - Mg0011 152, Sapporo
  - Mg0011 144, Sendai
  - Mg0011 163, Shinjuku-ku
  - Mg0011 141, Tokyo
- Norway (2):
  - Mg0011 140, Bergen
  - Mg0011 143, Oslo
- Poland (11):
  - Mg0011 195, Katowice
  - Mg0011 213, Katowice
  - Mg0011 192, Krakow
  - Mg0011 193, Krakow
  - Mg0011 211, Krakow
  - Mg0011 214, Lodz
  - Mg0011 205, Lublin
  - Mg0011 194, Nowa Sól
  - Mg0011 209, Poznan
  - Mg0011 201, Warsaw
  - Mg0011 210, Zabrze
- Spain (3):
  - Mg0011 133, Barcelona
  - Mg0011 168, Barcelona
  - Mg0011 138, Bilbao
- United Kingdom (2):
  - Mg0011 119, Oxford
  - Mg0011 130, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Weiss MD, Freimer M, Leite MI, Maniaol A, Utsugisawa K, Bloemers J, Boroojerdi B, Howard E, Savic N, Howard JF Jr. Improvement of fatigue in generalised myasthenia gravis with zilucoplan. J Neurol. 2024 May;271(5):2758-2767. doi: 10.1007/s00415-024-12209-3. Epub 2024 Feb 24. PMID 38400914
- [Result] de la Borderie G, Chimits D, Boroojerdi B, Brock M, Duda PW, Grimson F, Mahoney P, Strimenopoulou F, Cutter G, Aban I, Brauner S, Petersson M, Howard JF Jr, Bennett N. Maintenance of zilucoplan efficacy in patients with generalised myasthenia gravis up to 24 weeks: a model-informed analysis. Ther Adv Neurol Disord. 2024 Sep 21;17:17562864241279125. doi: 10.1177/17562864241279125. eCollection 2024. PMID 39314260
- [Result] Hewamadduma C, Freimer M, Genge A, Leite MI, Utsugisawa K, Vu T, Boroojerdi B, Grimson F, Savic N, Vanderkelen M, Howard JF Jr; RAISE-XT study team. Changes in corticosteroid and non-steroidal immunosuppressive therapy with long-term zilucoplan treatment in generalized myasthenia gravis. J Neurol. 2025 Jun 12;272(7):457. doi: 10.1007/s00415-025-13113-0. PMID 40504283
- [Derived] Howard JF Jr, Bresch S, Farmakidis C, Freimer M, Genge A, Hewamadduma C, Hinton J, Hussain Y, Juntas-Morales R, Kaminski HJ, Maniaol A, Mantegazza R, Masuda M, Nowak RJ, Sivakumar K, Smilowski M, Utsugisawa K, Vu T, Weiss MD, Zajda M, Bloemers J, Boroojerdi B, Brock M, de la Borderie G, Duda PW, Vanderkelen M, Leite MI; RAISE-XT Study Team*. Long-term safety and efficacy of zilucoplan in patients with generalized myasthenia gravis: interim analysis of the RAISE-XT open-label extension study. Ther Adv Neurol Disord. 2024 Apr 17;17:17562864241243186. doi: 10.1177/17562864241243186. eCollection 2024. PMID 38638673
- [Derived] Howard JF Jr, Bresch S, Genge A, Hewamadduma C, Hinton J, Hussain Y, Juntas-Morales R, Kaminski HJ, Maniaol A, Mantegazza R, Masuda M, Sivakumar K, Smilowski M, Utsugisawa K, Vu T, Weiss MD, Zajda M, Boroojerdi B, Brock M, de la Borderie G, Duda PW, Lowcock R, Vanderkelen M, Leite MI; RAISE Study Team. Safety and efficacy of zilucoplan in patients with generalised myasthenia gravis (RAISE): a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Neurol. 2023 May;22(5):395-406. doi: 10.1016/S1474-4422(23)00080-7. PMID 37059508